CLINICAL TRIAL: NCT03371316
Title: Preliminary Investigation of ViaShield™ Amnion Patch as an Anti-Adhesive Barrier in Hemicraniectomies
Acronym: ViaShield
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Site is no longer participating in study
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGC17-001
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Hemicraniectomies

STUDY DESIGN:
Intervention Model Description: All patients requiring a hemicraniectomy will also receive the amnion patch as an anti-adhesive barrier
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemicraniectomy Surgery with Viashield (Experimental): All patients requiring a hemicraniectomy surgery will receive the anti-adhesion barrier of amnion patch.
  Interventions: Biological: ViaShield

INTERVENTIONS:
Biological: ViaShield — Anti-adhesion scores using amnion patch

SUMMARY:
The goal of this study is to demonstrate that ViaShield™ amnion patch is effective in preventing fibroblast activity and hence soft tissue adhesions after a hemicraniectomy.

DETAILED DESCRIPTION:
A hemicraniectomy is a surgical procedure in which part of the skull is temporarily removed to relieve pressure on the underlying brain. Hemicraniectomies are typically performed on patients experiencing severe brain injury, usually due to stroke or trauma. In these cases, the brain injury and swelling is so severe that it can lead to brain compression and brain death. As a result, a surgeon will remove the bone flap to help with brain swelling and increased intracranial pressure. After the patient heals, a cranioplasty will be performed to restore the bone flap to its original location.

When the central nervous system is deprived of its normal covering, as is the case with hemicraniectomies, the exposed area becomes the site of cellular reaction from surrounding tissue1 and soft tissue adhesions frequently develop between the skin flap and the dura mater or exposed brain, which may lead to less than optimal clinical outcome.

ViaShield™ is an amnion patch produced from human amniotic membrane. Because of its inherent anti-adhesive properties, amnion serves as an ideal barrier against scarring and soft tissue adhesions to the neural elements, anterior vessels and hardware.

ELIGIBILITY:
Inclusion Criteria:

18 years of age minimum Informed consent signed by patient or next of kin

Exclusion Criteria:

Immunosuppressive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Adhesion | 4-8 months
  Adhesion tenacity scores post hemicraniectomies 0 No adhesions
  1. Thin membranous adhesions, no vessel attachment
  2. Mild adhesions, blunt dissection required
  3. Moderate adhesions, some sharp dissection required
  4. Tenacious adhesions, sharp instrument dissection required, vessels attached The lower the score the better the outcome for the patient

SECONDARY OUTCOMES:
Infections | From time of surgery to 8 months post-operative
  Wound Infections in or around hemicraniectomy site
hydrocephalus | From time of surgery to 8 months post-operative
  Accumulation of fluid around the brain

IPD SHARING:
Plan to Share IPD: No